CLINICAL TRIAL: NCT03177616
Title: Integrative Migraine Pain Alleviation Through Chiropractic Therapy
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: Brigham and Women's Hospital (Other); Palmer Center for Chiropractic Research (PCCR) (Other)
Responsible Party: Principal Investigator, Peter Wayne, Associate Professor of Medicine, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P000087
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Migraine; Migraine Disorders; Migraine With Aura; Migraine Without Aura; Migraine, Classic
Keywords: Migraine; Women; Adult; Feasibility; Safety; Pilot Randomized Trial; Randomized Control Trial; Chiropractic
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Subjects randomized to the usual care control group will continue using their usual medical care as prescribed by their physician. They are not to use any chiropractic treatment or begin new therapies.
- Chiropractic Treatment + Usual Care (Experimental): Patients will receive a course of 10 chiropractic treatments over a 14 week period. They are to also maintain their usual medical care as prescribed by their physician, but are not to begin any new therapies.
  Interventions: Other: Chiropractic Treatment

INTERVENTIONS:
Other: Chiropractic Treatment — The treatment plan will be customized to the patient's needs. The chiropractic interventions are summarized as follows:
  * posture correction/spinal stabilization exercises
  * soft tissue relaxation techniques
  * spinal manipulation (i.e. chiropractic adjustment)/mobilization
  * breathing and relaxing techniques
  * stretches, self-care
  * ergonomic modifications
  * bracing and supports
  Arms: Chiropractic Treatment + Usual Care

SUMMARY:
This pilot study evaluates the addition of chiropractic treatment to conventional neurological care in the treatment of migraine headaches in adult women. Half of the participants will receive 10 chiropractic treatments in addition to their usual care over a 14 week period, while the other half will continue their usual medical care alone, as prescribed by their physician during that time period.

DETAILED DESCRIPTION:
Chiropractic care is a commonly used therapeutic intervention for the treatment of pain disorders, and some smaller studies have shown that it might be helpful for migraines. This pilot study will use a comprehensive model of chiropractic treatment which can include soft tissue mobilization, spinal manipulation, and postural and spinal stabilization and correctional exercises.

Specific Aims:

Aim #1 - Determine the feasibility of conducting a randomized control trial (RCT) of chiropractic care in adult women with migraine.

Aim #2 - To provide preliminary data on the safety and effectiveness of chiropractic care on migraine frequency, severity, duration, and medication use in adult women with migraine.

Aim #3 - To provide preliminary estimates of the effects of chiropractic on disability, health-related quality of life, and psychosocial well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of episodic migraine with or without aura (International Classification of Headache Disorders-II)
* 4 to 13 days with migraines/month
* More than one year of migraines
* Agreeable to participate, commit to all study procedures, and to be randomized to either group
* Fluent in English (required to complete self-report instruments)

Exclusion Criteria:

* Currently, or having received chiropractic care in past 3 months for any condition
* Any major systemic illness or unstable medical or psychiatric condition (e.g. Parkinson's disease, cancer) requiring immediate treatment or that could lead to difficulty complying with the protocol
* History of stroke, carotid artery dissection, or vertebral artery dissection
* Head or neck trauma within the past year
* Diagnosis of medication overuse headache (International Classification of Headache Disorders-II)
* Began use of new prophylactic medication for migraine headaches within the last 3 months
* Currently taking prophylactic migraine medications other than propranolol and topiramate
* Failure to complete baseline diary recordings of migraine activity and medication use during run-in phase
* Currently, or having received Botox treatment for migraine
* Current alcohol or substance abuse (self-reported)
* Diagnosis of Ehlers-Danlos Syndrome

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the last four weeks of the intervention period in the number of migraine days. | From the baseline period to week 11 through week 14.
  Participants will record number of migraines experienced in provided logs.

SECONDARY OUTCOMES:
Changes from baseline to the post-intervention period in the number of migraine days. | From the baseline period to week 15 through week 18.
  Participants will record number of migraines experienced in provided logs for four weeks post-intervention.
Number of responders | From the baseline period to week 11 through week 14 and to week 15 through week 18.
  Participants who had a greater than 50% reduction in days with migraine per four week period.
Change from baseline in the severity of migraine | From the baseline period to week 11 through week 14 and to week 15 through week 18.
  Participants will record the severity of migraines on a scale of 1 to 10 in provided logs.
Change from baseline in the duration of migraine | From the baseline period to week 11 through week 14 and to week 15 through week 18.
  Participants will record the duration (hours) of migraines in provided logs.
Change from baseline in the doses of acute migraine medications used | From the baseline period to week 11 through week 14 and to week 15 through week 18.
  Participants will record the medications taken to treat/prevent their migraines in provided logs.
Change from baseline in the scores on the Headache Impact Test (HIT-6) questionnaire | From baseline to 14 weeks and 18 weeks
  The HIT-6 questionnaire evaluates headache related disability.
Change from baseline in the scores on the Migraine Disability Assessment (MIDAS) | From baseline to 14 weeks and 18 weeks
  The MIDAS is a 5-item questionnaire used to assess disability in migraine research.
Change from baseline in the Migraine Specific Quality of Life Questionnaire version 2.1 (MSQv2.1) | From baseline to 14 weeks and 18 weeks
  The MSQv2.1 measures how migraines affect a patient's daily life.
Change from baseline in Numeric Rating Pain Scale (NRS) | From baseline to 14 weeks and 18 weeks
  The NRS tool will be used to measure neck pain on a scale from 1 to 10.
Change from baseline in 9-item Patient Health Questionnaire (PHQ-9) | From baseline to 14 weeks and 18 weeks
  The PHQ-9 will be used to measure changes in mood.
Change from baseline in the Generalized Anxiety Disorder 7-item (GAD-7) | From baseline to 14 weeks and 18 weeks
  The GAD-7 will be used to measure changes in mood.
Change from baseline in the Patient Reported Outcome Measures Information System -29 item questionnaire (PROMIS-29) | From baseline to 14 weeks and 18 weeks
  The PROMIS-29 will be used to measure changes in mood.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wayne, Ph.D., Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- The Osher Clinical Center for Integrative Medicine at Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rist PM, Bernstein C, Kowalski M, Osypiuk K, Connor JP, Vining R, Long CR, Macklin EA, Wayne PM. Multimodal chiropractic care for migraine: A pilot randomized controlled trial. Cephalalgia. 2021 Mar;41(3):318-328. doi: 10.1177/0333102420963844. Epub 2020 Oct 13. PMID 33050719